CLINICAL TRIAL: NCT02177708
Title: Quantitative Determination of Brain Water Content in Patients During and After Hepatic Encepalopathy Measured by MR
Brief Title: Quantitative Determination of Brain Water Content in Patients During and After Hepatic Encepalopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Gitte Dam, MD, PHD, University of Aarhus
Other Study IDs: 34781
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Last update posted 2014-06-30 (Estimated); Status verified 2014-06

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
There is increasing evidence that the pathophysiology of hepatic encephalopathy (HE) is tightly associated with low-grade cerebral edema. Uptake of ammonia in astrocytes leads to osmotic swelling caused by glutamine formation. Previous studies were performed in covert HE patients or used indirect methods.

Methods: The investigators wish to describes quantitative measurement of localized water content using MRI water mapping in a cohort of patients with cirrhosis during an episode of overt HE type C and again after recovery. Furthermore patients with cirrhosis and no history of HE and healthy subjects will be investigated as controls.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type C HE during and after HE,
* Patients with stable cirrhosis and
* Healthy subjects

Exclusion Criteria:

* Patients with pace-maker
* Metal implants

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Type C HE
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Absolute brain water content measured by water mapping | Patients are recruited during an episode of acute HE, the patients are rescanned within a time frame of 6 weeks. Patients with stable cirrhosis and healthy subjects are scanned only once.

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Dam, MD, Phd, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus, Denmark